CLINICAL TRIAL: NCT05548374
Title: The Safety and Efficacy of Acupuncture in Moderate to Severe Cyclic Breast Pain
Brief Title: Acupuncture for Breast Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Yuanjie Sun, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-007-KY
Record Dates: First submitted 2022-09-13; First posted 2022-09-21 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Acupuncture; Mastodynia
Keywords: Chronic Breast Pain; Female
MeSH Terms: conditions — Mastodynia | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupucnture (Experimental): Treatment will start 2 weeks before the onset of menstruation in 3 consecutive menstrual cycles, three sessions per week (ideally every other day) in the first two menstrual cycles and two sessions per week in the last menstrual cycle, 16 sessions in total.
  Interventions: Device: Acupuncture
- Sham Acupuncture (Sham Comparator): Treatment will start 2 weeks before the onset of menstruation in 3 consecutive menstrual cycles, three sessions per week (ideally every other day) in the first two menstrual cycles and two sessions per week in the last menstrual cycle, 16 sessions in total.
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: Acupuncture — The acupoints of Shangyintang, Danzhong(RNl7), Jvque(RN14), Liangmen(ST21), Zhongwan(RNl2), Hegu(LI4), Waiguan(SJ5), Zusanli(ST36), Sanyinjiao(SP6), Taichong(LR3) are selected as main acupoints and used per treatment. The other three acupoints will be chosen one each session according to the syndrome differentiation: Taixi (KI3) for liver and kidney deficiency, Fenglong (ST40) for spleen deficiency and phlegm coagulation, and Xuehai (SP10) for qi-stagnation and blood-stasis. Sterile adhesive pads will be placed on the acupoints after skin disinfection. Hwato-brand disposable acupuncture needles (size 0.30×40mm) will be inserted into the acupoints through the adhesive pads. Afterwards, the acupuncture will be lifted, thrusted and twirled gently for 3 times to achieve deqi sensation and manipulated every ten minutes during 30-minute maintenance.
  Arms: Acupucnture
Device: Sham acupuncture — The acupoints of Shangyintang, Danzhong(RNl7), Jvque(RN14), Liangmen(ST21), Zhongwan(RNl2), Hegu(LI4), Waiguan(SJ5), Zusanli(ST36), Sanyinjiao(SP6), Taichong(LR3) are selected as main acupoints and used per treatment. The other three acupoints will be chosen one each session according to the syndrome differentiation: Taixi (KI3) for liver and kidney deficiency, Fenglong (ST40) for spleen deficiency and phlegm coagulation, and Xuehai (SP10) for qi-stagnation and blood-stasis. Sterile adhesive pads will be placed on the acupoints after skin disinfection. The needles (with the handle identical to the needles in the acupuncture group and the body at a size 0.30 × 25 mm) will be inserted into adhesive pads without skin penetration. Needles will be lifted, thrusted and twirled gently for 3 times to mimic real acupuncture. No manipulation will be conducted during 30-minute maintenance.
  Arms: Sham Acupuncture

SUMMARY:
This study is conducted to assess the efficacy and safety of acupuncture in moderate to severe cyclic breast pain.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the diagnosis criteria of cyclic breast pain.
* Female patients aged between 18 and 55.
* Relatively regular menstrual cycle.
* Cyclic breast pain lasting for 3 consecutive menstrual cycles or more.
* The score of worst pain ≥5 on Numerical Rating Scale and any level of breast pain lasting 5-21 days during the run-in period of one menstrual cycle.
* No previous experience of acupuncture for breast diseases.
* Willing to use nonhormonal contraceptives if any risk of pregnancy.
* Volunteer to the trial and signing written informed consent.

Exclusion Criteria:

* Noncyclic breast pain.
* Extramammary pain only.
* A history of breast cancer or suspicious of malignancy breast disease by examinations.
* The Breast Imaging Reporting and Data System (BI-RADS) category 4-6 in ultrasound or mammography examinations.
* Combined with mastitis.
* Breast pain following injury, surgery, hormones, and/or other drugs.
* Usage of hormones (including hormonal contraceptives) in the past three months.
* Combined with severe diseases in the cardiac, respiratory, renal, liver, and hematopoietic systems, psychiatric disorder and/or cognitive disorders.
* A history of bilateral ovariectomy or premature ovarian failure.
* Pregnancy, lactation, or wishing to conceive before the end of the trial.
* Poor adherence.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
The change from baseline in the numerical rating scale (NRS) score on the worst breast pain. | Through the Cycle 3 (each cycle is 25-35 days)
  Participants will fill in the Cardiff Breast Pain Chart to assess the intensity of worst and average pain daily in the form of NRS score ranging from 0-10. 0 refers to no pain and 10 refers to the worst pain imaginable. The highest NRS score on the worst breast pain during the cycle is defined as the final score on the worst pain.

SECONDARY OUTCOMES:
The change from baseline in the numerical rating scale (NRS) score on the worst breast pain. | Through the Cycle 1, Cycle 2, Cycle 6 and Cycle 9 (each cycle is 25-35 days)
  Participants will fill in the Cardiff Breast Pain Chart to assess the intensity of worst and average pain daily in the form of NRS score ranging from 0-10. 0 refers to no pain and 10 refers to the worst pain imaginable. The highest NRS score on the worst breast pain during the cycle is defined as the final score on the worst pain.
The change from baseline in the numerical rating scale (NRS) score on the average breast pain. | Through the Cycle 1, Cycle 2, Cycle 3, Cycle 6 and Cycle 9 (each cycle is 25-35 days)
  Participants will fill in the Cardiff Breast Pain Chart to assess the intensity of worst and average pain daily in the form of NRS score ranging from 0-10. 0 refers to no pain and 10 refers to the worst pain imaginable. The average NRS score on the average breast pain during the cycle is defined as the mean of the average pain score during the cycle.
Proportion of participants with at least 50% reduction of NRS score on the worst breast pain. | Through the Cycle 1, Cycle 2, Cycle 3, Cycle 6 and Cycle 9 (each cycle is 25-35 days)
  Participants will fill in the Cardiff Breast Pain Chart to assess the intensity of worst and average pain daily in the form of NRS score ranging from 0-10. 0 refers to no pain and 10 refers to the worst pain imaginable. The highest NRS score on the worst breast pain during the cycle is defined as the final score on the worst pain.
Proportion of participants with at least 50% reduction of NRS score on the average breast pain. | Through the Cycle 1, Cycle 2, Cycle 3, Cycle 6 and Cycle 9 (each cycle is 25-35 days)
  Participants will fill in the Cardiff Breast Pain Chart to assess the intensity of worst and average pain daily in the form of NRS score ranging from 0-10. 0 refers to no pain and 10 refers to the worst pain imaginable. The average NRS score on the average breast pain during the cycle is defined as the mean of the average pain score during the cycle.
The change from baseline in the number of days with a NRS score of 5 or over on the worst breast pain. | Through the Cycle 1, Cycle 2, Cycle 3, Cycle 6 and Cycle 9 (each cycle is 25-35 days)
  Participants will fill in the Cardiff Breast Pain Chart to assess the intensity of worst and average pain daily in the form of NRS score ranging from 0-10. 0 refers to no pain and 10 refers to the worst pain imaginable. The highest NRS score on the worst breast pain during the cycle is defined as the final score on the worst pain.
The change from baseline in the number of days with breast pain. | Through the Cycle 1, Cycle 2, Cycle 3, Cycle 6 and Cycle 9 (each cycle is 25-35 days)
  Participants will fill in the Cardiff Breast Pain Chart to assess the intensity of worst and average pain daily in the form of NRS score ranging from 0-10. 0 refers to no pain and 10 refers to the worst pain imaginable.
The proportion of patients reported "very much improved" or "much improved" per the Patient Global Impression of Change (PGIC). | At the end of the Cycle 3, Cycle 6 and Cycle 9 (each cycle is 25-35 days)
  PGIC is a 7-point scale reflecting patient's self-rating of overall improvement: "very much improved", "much improved", "minimally improved", "no change", "minimally worse", "much worse" or "very much worse".
The impact of breast pain on sexual life, daily life, mood and sleep rated by NRS scale. | At the end of the Cycle 1, Cycle 2, Cycle 3, Cycle 6 and Cycle 9 (each cycle is 25-35 days)
  NRS ranges from 0 to 10, with 0 indicating no impact and 10 indicating influence completely, and higher scores represent severer impact.
The change from baseline in the Sort Form 12-item Health Survey (SF-12). | At the end of the Cycle 1, Cycle 2, Cycle 3, Cycle 6 and Cycle 9 (each cycle is 25-35 days)
  The SF-12 is a general health questionnaire consisting of 12 questions. It investigates the patient's state of health via 8 different dimensions of general health perception, physical health, limited physical role function, physical pain, vitality, mental health, limited emotional role function, and social functioning. The sores of SF-12 range from 0 to 100, with higher scores indicating better physical and mental health functioning.
The change from baseline in the total and sub scores of Hospital Anxiety and Depression Scale (HADS). | At the end of the Cycle 1, Cycle 2, Cycle 3, Cycle 6 and Cycle 9 (each cycle is 25-35 days)
  HADS consists of 14 items, which are divided into two 7-item subscales to reflect a state of generalized anxiety and the depression. The respondent rates each item on a 4-point scale ranging from 0 (absence) to 3 (extreme presence). The total scores of HADS ranges from 0 to 42, with higher scores indicating severer symptoms.

OTHER OUTCOMES:
Expectance assessment | At the end of Cycle 0 (each cycle is 25-35 days)
  Patients will be asked what do you think the condition of breast pain will be in three menstrual cycles.
Assessment of belief in acupuncture | At the end of the Cycle 0 and Cycle 3 (each cycle is 25-35 days)
  Patients will be asked do you think acupuncture can help to treat your breast pain.
Blinding assessment | Within 5 minutes after the last treatment
  Participants will be ask do you think you have received traditional acupuncture in the past 3 menstrual cycles.
Adherence assessment | Through the Cycle 1, cycle 2, and cycle 3 (each cycle is 25-35 days)
  Adherence will be assessed via counting treatment sessions. Those complete over 80% treatment sessions will be defined as of good adherence.
Proportion of participants using rescue medicine. | Through study completion, an average of one and a half years.
Proportion of participants using concomitant medicine or therapy that might impact breast pain. | Through study completion, an average of one and a half years.

CONTACTS AND LOCATIONS:
Locations (1):
- Yuanjie Sun, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data and data dictionary will be available with publication until six months after publication.
  Formal request should be sent to puzhisun@163.com with a methodologically sound proposal.
  Researchers whose proposal has been approved will sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available with publication until six months after publication.
Access Criteria: Formal request should be sent to puzhisun@163.com with a methodologically sound proposal. Researchers whose proposal has been approved will sign a data access agreement.